CLINICAL TRIAL: NCT01349309
Title: The Effect of Prophylactic Swallowing Exercises on Head and Neck Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GCO # 07-0462
Record Dates: First submitted 2011-02-28; First posted 2011-05-06 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-12

CONDITIONS: Dysphagia
Keywords: Prophylactic Swallowing Exercises; Head and Neck Cancer; Dysphagia
MeSH Terms: conditions — Deglutition Disorders; Head and Neck Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Swallowing Exercise Group (Experimental): Swallowing Exercise Group: This arm will undergo the protocol that involves intensive swallowing exercises to begin at the start of the cancer treatment. Those patients randomized to the intensive therapy protocol will be required to participate in weekly swallowing therapy sessions either in person or over the phone and perform the learned swallowing exercises three times a day. In addition, these patients will document their swallowing practice on a daily basis.
  Interventions: Behavioral: Swallowing Exercise Group
- Control (No Intervention): Control Arm: This arm will receive the standard of care which provides swallowing evaluation and treatment once symptoms of swallowing dysfunction are experienced by the patient.

INTERVENTIONS:
Behavioral: Swallowing Exercise Group — Swallowing Exercises
  Perform each exercise 10 times. Do these 3 times a day. Vary the order of the exercises.
  Effortful Swallow: As you swallow squeeze hard with all your muscles. (Can do with water or without)
  Super Supraglottic Swallow:
  Inhale and hold your breath very tightly, bearing down. Keep holding your breath and bearing down as you swallow. Cough when you are finished. (Can do with water or without)
  Tongue Hold Maneuver:
  Gently hold your tongue in between your front teeth and swallow your saliva.
  Tongue Retraction:
  Pull the back of your tongue to the back of your mouth and hold.
  Mendelsohn Maneuver:
  Swallow your saliva and pay attention to your neck as you swallow. Try to feel that something (your Adam's apple of voice box) lifts and lowers as you swallow. Now, when you swallow and you feel something lift as you swallow don't let it drop. Hold it with your muscles for several seconds.
  Other Names: Prophylactic Swallowing Exercises
  Arms: Swallowing Exercise Group

SUMMARY:
The purpose of this study is to find out if doing prophylactic or preventative swallowing exercises from the start of cancer treatment can improve the ability to swallow when the treatment is completed and beyond.

DETAILED DESCRIPTION:
Study Type: Prospective Randomized Clinical Trial

Introduction:

Organ sparing treatment for advanced head and neck cancer can affect the swallowing mechanism via fibrosis of the structures responsible for effective and efficient bolus movement from the oral cavity and through the pharynx into the esophagus. This fibrosis may result in significant impairment of bolus transport. Range of motion exercises for the swallowing structures may decrease the fibrotic effects of the radiation treatment and improve swallowing outcomes after treatment.

Intervention:

Patients who have been diagnosed with head and neck cancer and who will be receiving radiation therapy either with or without chemotherapy as cancer treatment will be randomized to one of two swallowing treatment protocols. The first protocol will include the initiation of intensive swallowing exercises to begin at the start of the cancer treatment. The second treatment protocol will include the standard of care which provides swallowing evaluation and treatment once symptoms of swallowing dysfunction are experienced by the patient. Patients will not be given a choice of swallowing protocol. Those patients randomized to the intensive therapy protocol will be required to participate in weekly swallowing therapy sessions either in person or over the phone and perform the learned swallowing exercises three times a day. In addition, these patients will document their swallowing practice on a daily basis. The same investigator will provide all the swallowing treatment assuring that all patients get the same treatment approach.

All patients will fill out a questionnaire about their swallowing ability called the Performance Status Scale for Head and Neck Cancer Patients (PSS-H&N). This is a quick, clinician rated instrument consisting of three subscales: normalcy of diet, public eating and intelligibility of speech. This scale has been proven reliable across raters and sensitive to functional differences across a broad spectrum of head and neck cancer patients. This questionnaire will be completed at the start of the cancer treatment, at the completion of the treatment and at 3, 6, 12 and 24 months after treatment. In addition, the nature of the patient's oral intake will be documented by the investigator using the Functional Oral Intake Scale (FOIS) which is a seven point scale of diet tolerance. This will be performed at the same intervals as the PSS-H&N. Presence or absence of PEG feedings will also be documented at these same times. These scales will then be used to compare the swallowing outcomes of the patients in the two different treatment protocols.

ELIGIBILITY:
Inclusion criteria:

* Patient diagnosed with head and neck cancer who will be receiving radiation therapy either alone of with chemotherapy as their treatment modality.

Exclusion criteria:

* Patients with a history of neurologic disease
* Patients with previous head and neck cancer or surgical or radiation treatment to the head and neck region
* Patients taking medication that might effect their swallowing function
* Patients with gastroenterologic dysfunction
* Patients who have previously undergone swallowing therapy
* Patients with cognitive impairments that limit their ability to follow and comply with multi-step commands

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2007-06; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Performance Status Scale for Head and Neck Cancer Patients and Functional Oral Intake Scale (PSS-H&N). | This will be completed at the start of the cancer treatment. Participants will be followed for up to 24 months after treatment.
  This is a quick, clinician rated instrument consisting of three subscales: normalcy of diet, public eating and intelligibility of speech. This scale has been proven reliable across raters and sensitive to functional differences across a broad spectrum of head and neck cancer patients. The Performance Status Scale for Head and Neck Cancer Patients (PSS-H&N) questionnaire will be completed at the start of the cancer treatment, at the completion of the treatment and at 3, 6, 12 and 24 months after treatment.
Performance Status Scale for Head and Neck Cancer Patients and Functional Oral Intake Scale (PSS-H&N). | This will be completed at the completion of treatment. Participants will be followed for up to 24 months after treatment.
  This is a quick, clinician rated instrument consisting of three subscales: normalcy of diet, public eating and intelligibility of speech. This scale has been proven reliable across raters and sensitive to functional differences across a broad spectrum of head and neck cancer patients. The Performance Status Scale for Head and Neck Cancer Patients (PSS-H&N) questionnaire will be completed at the start of the cancer treatment, at the completion of the treatment and at 3, 6, 12 and 24 months after treatment.
Performance Status Scale for Head and Neck Cancer Patients and Functional Oral Intake Scale (PSS-H&N). | This will be completed at 3 months post treatment. Participants will be followed for up to 24 months after treatment.
  This is a quick, clinician rated instrument consisting of three subscales: normalcy of diet, public eating and intelligibility of speech. This scale has been proven reliable across raters and sensitive to functional differences across a broad spectrum of head and neck cancer patients. The Performance Status Scale for Head and Neck Cancer Patients (PSS-H&N) questionnaire will be completed at the start of the cancer treatment, at the completion of the treatment and at 3, 6, 12 and 24 months after treatment.
Performance Status Scale for Head and Neck Cancer Patients and Functional Oral Intake Scale (PSS-H&N). | This will be completed at 6 months post treatment. Participants will be followed for up to 24 months after treatment.
  This is a quick, clinician rated instrument consisting of three subscales: normalcy of diet, public eating and intelligibility of speech. This scale has been proven reliable across raters and sensitive to functional differences across a broad spectrum of head and neck cancer patients. The Performance Status Scale for Head and Neck Cancer Patients (PSS-H&N) questionnaire will be completed at the start of the cancer treatment, at the completion of the treatment and at 3, 6, 12 and 24 months after treatment.
Performance Status Scale for Head and Neck Cancer Patients and Functional Oral Intake Scale (PSS-H&N). | This will be completed at 12 months post treatment. Participants will be followed for up to 24 months after treatment.
  This is a quick, clinician rated instrument consisting of three subscales: normalcy of diet, public eating and intelligibility of speech. This scale has been proven reliable across raters and sensitive to functional differences across a broad spectrum of head and neck cancer patients. The Performance Status Scale for Head and Neck Cancer Patients (PSS-H&N) questionnaire will be completed at the start of the cancer treatment, at the completion of the treatment and at 3, 6, 12 and 24 months after treatment.
Performance Status Scale for Head and Neck Cancer Patients and Functional Oral Intake Scale (PSS-H&N). | This will be completed at 24 months post treatment. Participants will be followed for up to 24 months after treatment.
  This is a quick, clinician rated instrument consisting of three subscales: normalcy of diet, public eating and intelligibility of speech. This scale has been proven reliable across raters and sensitive to functional differences across a broad spectrum of head and neck cancer patients. The Performance Status Scale for Head and Neck Cancer Patients (PSS-H&N) questionnaire will be completed at the start of the cancer treatment, at the completion of the treatment and at 3, 6, 12 and 24 months after treatment.
Functional Oral Intake Scale (FOIS) | This will be completed at the start of the cancer treatment. Participants will be followed for up to 24 months after treatment.
  A seven point scale of diet tolerance.
Functional Oral Intake Scale (FOIS) | This will be completed at the completion of treatment. Participants will be followed for up to 24 months after treatment.
  A seven point scale of diet tolerance.
Functional Oral Intake Scale (FOIS) | This will be completed at 3 post treatment. Participants will be followed for up to 24 months after treatment.
  A seven point scale of diet tolerance.
Functional Oral Intake Scale (FOIS) | This will be completed at 6 months post treatment. Participants will be followed for up to 24 months after treatment.
  A seven point scale of diet tolerance.
Functional Oral Intake Scale (FOIS) | This will be completed at 12 months post treatment. Participants will be followed for up to 24 months after treatment.
  A seven point scale of diet tolerance.
Functional Oral Intake Scale (FOIS) | This will be completed at 24 months post treatment. Participants will be followed for up to 24 months after treatment.
  A seven point scale of diet tolerance.

CONTACTS AND LOCATIONS:
Overall Officials: Tamar Kotz, MS, CCC, SLP, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Background] Lee NY, de Arruda FF, Puri DR, Wolden SL, Narayana A, Mechalakos J, Venkatraman ES, Kraus D, Shaha A, Shah JP, Pfister DG, Zelefsky MJ. A comparison of intensity-modulated radiation therapy and concomitant boost radiotherapy in the setting of concurrent chemotherapy for locally advanced oropharyngeal carcinoma. Int J Radiat Oncol Biol Phys. 2006 Nov 15;66(4):966-74. doi: 10.1016/j.ijrobp.2006.06.040. PMID 17145527
- [Background] El-Sayed S, Nelson N. Adjuvant and adjunctive chemotherapy in the management of squamous cell carcinoma of the head and neck region. A meta-analysis of prospective and randomized trials. J Clin Oncol. 1996 Mar;14(3):838-47. doi: 10.1200/JCO.1996.14.3.838. PMID 8622032
- [Background] Pignon JP, Bourhis J, Domenge C, Designe L. Chemotherapy added to locoregional treatment for head and neck squamous-cell carcinoma: three meta-analyses of updated individual data. MACH-NC Collaborative Group. Meta-Analysis of Chemotherapy on Head and Neck Cancer. Lancet. 2000 Mar 18;355(9208):949-55. PMID 10768432
- [Background] Mendenhall WM, Amdur RJ, Stringer SP, Villaret DB, Cassisi NJ. Radiation therapy for squamous cell carcinoma of the tonsillar region: a preferred alternative to surgery? J Clin Oncol. 2000 Jun;18(11):2219-25. doi: 10.1200/JCO.2000.18.11.2219. PMID 10829041
- [Background] Kramer S, Gelber RD, Snow JB, Marcial VA, Lowry LD, Davis LW, Chandler R. Combined radiation therapy and surgery in the management of advanced head and neck cancer: final report of study 73-03 of the Radiation Therapy Oncology Group. Head Neck Surg. 1987 Sep-Oct;10(1):19-30. doi: 10.1002/hed.2890100105. PMID 3449477
- [Background] Robbins KT. Barriers to winning the battle with head-and-neck cancer. Int J Radiat Oncol Biol Phys. 2002 May 1;53(1):4-5. doi: 10.1016/s0360-3016(02)02713-x. No abstract available. PMID 12007934
- [Background] Calais G, Alfonsi M, Bardet E, Sire C, Germain T, Bergerot P, Rhein B, Tortochaux J, Oudinot P, Bertrand P. Randomized trial of radiation therapy versus concomitant chemotherapy and radiation therapy for advanced-stage oropharynx carcinoma. J Natl Cancer Inst. 1999 Dec 15;91(24):2081-6. doi: 10.1093/jnci/91.24.2081. PMID 10601378
- [Background] Brizel DM, Albers ME, Fisher SR, Scher RL, Richtsmeier WJ, Hars V, George SL, Huang AT, Prosnitz LR. Hyperfractionated irradiation with or without concurrent chemotherapy for locally advanced head and neck cancer. N Engl J Med. 1998 Jun 18;338(25):1798-804. doi: 10.1056/NEJM199806183382503. PMID 9632446
- [Background] Vokes EE, Stenson K, Rosen FR, Kies MS, Rademaker AW, Witt ME, Brockstein BE, List MA, Fung BB, Portugal L, Mittal BB, Pelzer H, Weichselbaum RR, Haraf DJ. Weekly carboplatin and paclitaxel followed by concomitant paclitaxel, fluorouracil, and hydroxyurea chemoradiotherapy: curative and organ-preserving therapy for advanced head and neck cancer. J Clin Oncol. 2003 Jan 15;21(2):320-6. doi: 10.1200/JCO.2003.06.006. PMID 12525525
- [Background] Newman LA, Vieira F, Schwiezer V, Samant S, Murry T, Woodson G, Kumar P, Robbins KT. Eating and weight changes following chemoradiation therapy for advanced head and neck cancer. Arch Otolaryngol Head Neck Surg. 1998 May;124(5):589-92. doi: 10.1001/archotol.124.5.589. PMID 9604988
- [Background] Adelstein DJ, Saxton JP, Lavertu P, Rybicki LA, Esclamado RM, Wood BG, Strome M, Carroll MA. Maximizing local control and organ preservation in stage IV squamous cell head and neck cancer With hyperfractionated radiation and concurrent chemotherapy. J Clin Oncol. 2002 Mar 1;20(5):1405-10. doi: 10.1200/JCO.2002.20.5.1405. PMID 11870186
- [Background] Smith RV, Kotz T, Beitler JJ, Wadler S. Long-term swallowing problems after organ preservation therapy with concomitant radiation therapy and intravenous hydroxyurea: initial results. Arch Otolaryngol Head Neck Surg. 2000 Mar;126(3):384-9. doi: 10.1001/archotol.126.3.384. PMID 10722013
- [Background] Hutcheson KA, Barringer DA, Rosenthal DI, May AH, Roberts DB, Lewin JS. Swallowing outcomes after radiotherapy for laryngeal carcinoma. Arch Otolaryngol Head Neck Surg. 2008 Feb;134(2):178-83. doi: 10.1001/archoto.2007.33. PMID 18283161
- [Background] Bleier BS, Levine MS, Mick R, Rubesin SE, Sack SZ, McKinney K, Mirza N. Dysphagia after chemoradiation: analysis by modified barium swallow. Ann Otol Rhinol Laryngol. 2007 Nov;116(11):837-41. doi: 10.1177/000348940711601108. PMID 18074669
- [Background] Murry T, Madasu R, Martin A, Robbins KT. Acute and chronic changes in swallowing and quality of life following intraarterial chemoradiation for organ preservation in patients with advanced head and neck cancer. Head Neck. 1998 Jan;20(1):31-7. doi: 10.1002/(sici)1097-0347(199801)20:13.0.co;2-4. PMID 9464950
- [Background] Pauloski BR, Logemann JA. Impact of tongue base and posterior pharyngeal wall biomechanics on pharyngeal clearance in irradiated postsurgical oral and oropharyngeal cancer patients. Head Neck. 2000 Mar;22(2):120-31. doi: 10.1002/(sici)1097-0347(200003)22:23.0.co;2-u. PMID 10679899
- [Background] Kotz T, Costello R, Li Y, Posner MR. Swallowing dysfunction after chemoradiation for advanced squamous cell carcinoma of the head and neck. Head Neck. 2004 Apr;26(4):365-72. doi: 10.1002/hed.10385. PMID 15054740
- [Background] Eisbruch A, Lyden T, Bradford CR, Dawson LA, Haxer MJ, Miller AE, Teknos TN, Chepeha DB, Hogikyan ND, Terrell JE, Wolf GT. Objective assessment of swallowing dysfunction and aspiration after radiation concurrent with chemotherapy for head-and-neck cancer. Int J Radiat Oncol Biol Phys. 2002 May 1;53(1):23-8. doi: 10.1016/s0360-3016(02)02712-8. PMID 12007937
- [Background] Lazarus CL, Logemann JA, Pauloski BR, Colangelo LA, Kahrilas PJ, Mittal BB, Pierce M. Swallowing disorders in head and neck cancer patients treated with radiotherapy and adjuvant chemotherapy. Laryngoscope. 1996 Sep;106(9 Pt 1):1157-66. doi: 10.1097/00005537-199609000-00021. PMID 8822723
- [Background] Lazarus CL, Logemann JA, Pauloski BR, Rademaker AW, Larson CR, Mittal BB, Pierce M. Swallowing and tongue function following treatment for oral and oropharyngeal cancer. J Speech Lang Hear Res. 2000 Aug;43(4):1011-23. doi: 10.1044/jslhr.4304.1011. PMID 11386468
- [Background] Kotz T, Abraham S, Beitler JJ, Wadler S, Smith RV. Pharyngeal transport dysfunction consequent to an organ-sparing protocol. Arch Otolaryngol Head Neck Surg. 1999 Apr;125(4):410-3. doi: 10.1001/archotol.125.4.410. PMID 10208678
- [Background] Logemann JA, Pauloski BR, Rademaker AW, Colangelo LA. Super-supraglottic swallow in irradiated head and neck cancer patients. Head Neck. 1997 Sep;19(6):535-40. doi: 10.1002/(sici)1097-0347(199709)19:63.0.co;2-4. PMID 9278762
- [Background] Lazarus C, Logemann JA, Song CW, Rademaker AW, Kahrilas PJ. Effects of voluntary maneuvers on tongue base function for swallowing. Folia Phoniatr Logop. 2002 Jul-Aug;54(4):171-6. doi: 10.1159/000063192. PMID 12169803
- [Background] Lazarus C, Logemann JA, Gibbons P. Effects of maneuvers on swallowing function in a dysphagic oral cancer patient. Head Neck. 1993 Sep-Oct;15(5):419-24. doi: 10.1002/hed.2880150509. PMID 8407314
- [Background] Kulbersh BD, Rosenthal EL, McGrew BM, Duncan RD, McColloch NL, Carroll WR, Magnuson JS. Pretreatment, preoperative swallowing exercises may improve dysphagia quality of life. Laryngoscope. 2006 Jun;116(6):883-6. doi: 10.1097/01.mlg.0000217278.96901.fc. PMID 16735913
- [Background] Carroll WR, Locher JL, Canon CL, Bohannon IA, McColloch NL, Magnuson JS. Pretreatment swallowing exercises improve swallow function after chemoradiation. Laryngoscope. 2008 Jan;118(1):39-43. doi: 10.1097/MLG.0b013e31815659b0. PMID 17989581
- [Result] Kotz T, Federman AD, Kao J, Milman L, Packer S, Lopez-Prieto C, Forsythe K, Genden EM. Prophylactic swallowing exercises in patients with head and neck cancer undergoing chemoradiation: a randomized trial. Arch Otolaryngol Head Neck Surg. 2012 Apr;138(4):376-82. doi: 10.1001/archoto.2012.187. PMID 22508621